CLINICAL TRIAL: NCT03707717
Title: An Open-Label, Multicenter, Randomized, Parallel-Group, 3-Arm, Single-Dose Bioequivalence Study of Bimekizumab Injected Subcutaneously Either by a Prefilled Syringe or by an Auto-Injector in Adult Healthy Participants
Brief Title: A Study to Compare the Blood Level of Bimekizumab Injected Subcutaneously Either by a Prefilled Syringe or by an Auto-injector in Adult Healthy Volunteer Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UP0033; 2017-004403-48 (EudraCT Number)
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteers
Keywords: BKZ; UCB4940; Auto-Injector; Healthy Participants
MeSH Terms: interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bimekizumab-SS (Experimental): Subjects randomized to this arm will receive bimekizumab administered subcutaneously with a prefilled syringe.
  Interventions: Drug: Bimekizumab
- Bimekizumab-AI (Experimental): Subjects randomized to this arm will receive bimekizumab administered subcutaneously with an auto-injector.
  Interventions: Drug: Bimekizumab
- Bimekizumab-TN (Experimental): Subjects randomized to this arm will receive bimekizumab administered subcutaneously with a reference device.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive a pre-specified sequence of bimekzumab in the Treatment Period.
  Other Names: BKZ; UCB4940

SUMMARY:
The purpose of the study is to evaluate the pharmakokinetics (PK), safety, tolerability, and immunogenicity of bimekizumab (BKZ) when administered subcutaneously (sc) via 3 different BKZ delivery devices in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant is male or female aged >=18 years and <=55 years at Screening Visit
* Participant must be in good health (physically and mentally) as determined by the Investigator based on medical history (any chronic and acute illness), physical examination, vital signs, 12-lead electrocardiogram (ECG), and laboratory screening tests during the Screening Period
* Participant has a body mass index (BMI) of 18-32 kg/m2 and a minimum body weight of 50 kg for male participants and 45 kg for female participants, and a maximum body weight of 100 kg for all participants
* Participant is willing to abstain from alcohol-, tobacco-, and caffeine-containing products for 48 h prior to admission into the clinic and during the entire in-clinic stay

Exclusion Criteria:

* Subject has an active infection (except common cold), a serious infection, or a history of opportunistic, recurrent or chronic infections
* Participant has a history of a positive tuberculosis (TB) test or evidence of possible TB or latent TB infection at Screening Visit
* Participant has concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection
* Female participant who is pregnant, or plans to become pregnant during the study, or lactating, or sexually active with childbearing potential who is not using a medically accepted birth control method
* Participants receiving any live (includes attenuated) vaccination within the 8 weeks prior to Screening visit (eg, inactivated influenza and pneumococcal vaccines are allowed but nasal influenza vaccination is not permitted). Live vaccines are not allowed during the study or for 20 weeks after the last dose of the IMP
* Participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the participant's ability to participate in this study
* Participant has active neoplastic disease or history of neoplastic disease within 5 years of Screening Visit (except for basal or squamous cell carcinoma of the skin or carcinoma in situ that has been definitively treated with standard of care)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed bimekizumab (BKZ) plasma drug concentration (Cmax) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  The Cmax is the maximum plasma drug concentration of BKZ observed from pharmacokinetic samples taken at predefined time points.
Area under the BKZ plasma concentration-time curve from time zero to last quantifiable concentration (AUCt) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  The AUCt is the area under the plasma concentration-time curve from time zero to last quantifiable concentration (AUCt) of BKZ as determined using the linear trapezoidal rule.
Area under the BKZ plasma concentration-time curve from time zero to infinity (AUC) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  The area under the plasma concentration-time curve from time zero to infinity (AUC) of BKZ is calculated as AUC=AUCt+Clast/lambdaz, where Clast is the last quantifiable plasma concentration and λz is the apparent terminal elimination rate constant.
Percentage of subjects with at least one Adverse Event (AE) from first bimekizumab (BKZ) dose up to Safety Follow Up | From Baseline to Safety Follow Up (up to Day 140)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Percentage of subjects with at least one Serious Adverse Event (SAE) from first bimekizumab (BKZ) dose up to Safety Follow Up | From Baseline to Safety Follow Up (up to Day 140)
  A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is as infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above

SECONDARY OUTCOMES:
Percentage of the AUC extrapolated from the last quantifiable BKZ plasma concentration (%AUCex) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  The percentage of the AUC extrapolated from the last quantifiable BKZ plasma concentration (Clast) is computed from plasma concentrations of pharmacokinetic samples taken at predefined time points.
Time of occurrence of the maximum observed BKZ plasma drug concentration (tmax) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  Tmax is the time to reach maximum plasma concentration.
Apparent terminal half-life (t1/2) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  Apparent terminal half-life, reported in units of days, as determined via simple linear regression (slope=-lambdaz) of natural log (ln) concentration versus time for data points in the terminal phase of the concentration-time curve. t1/2 is calculated as ln2/lambdaz.
Apparent terminal elimination rate constant (lambdaz) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  The lambdaz is the rate constant of elimination.
Total body plasma clearance for BKZ (CL/F) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  The total body clearance (CL/F) for BKZ will be calculated as Dose/AUC. Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the plasma.
Volume of distribution for BKZ (Vz/F) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  Volume of distribution (Vz/F) for BKZ will be calculated as CL/lambdaz.
Time to last quantifiable BKZ plasma concentration (tmin) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  Tmin is the time to last quantifiable plasma concentration for BKZ.
Incidence of Anti-drug-antibodies (ADABs) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  Anti-drug-antibodies (ADABs) will be determined from blood samples taken at predefined timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (2):
- Up0033 002, Baltimore, Maryland, United States
- Up0033 001, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No